CLINICAL TRIAL: NCT03241108
Title: Randomized, Placebo-Controlled, Double Blind, Multicenter Phase 2 Study to Explore Tolerability, Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of Intravenous Multiple Infusions of NI-0101, an Anti-Toll Like Receptor 4 Monoclonal Antibody in Patients With Rheumatoid Arthritis
Brief Title: Study of an Anti-TLR4 mAb in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NI-0101-04; 2016-005017-45 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-08-07 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — NI-0101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NI-0101 (Experimental): A therapeutic humanized monoclonal antibody, administered by intravenous infusion every 2 weeks.
  Interventions: Drug: NI-0101
- Placebo (Placebo Comparator): The placebo matches NI-0101 without active ingredient, administered by intravenous infusion every 2 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NI-0101 — Humanized immunoglobulin gamma 1 (IgG1) kappa monoclonal antibody targeting TLR4
  Arms: NI-0101
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, PoC, randomized, placebo-controlled, double blind, international multicentre study to explore the effect of a new antibody to treat patients with Rheumatoid Arthritis

DETAILED DESCRIPTION:
The study foresees the randomization of at least 81 moderate to severe, ACPA positive, RA patients who are inadequate responders to MTX, in two double blind arms (NI-0101:placebo, with a ratio of 2:1). Patients will receive NI-0101 or placebo infusions up to a maximum of 6 administrations (every two weeks for 12 weeks). All patients will continue receiving a stable dose of MTX. After 12 weeks, patients will enter the follow up period with monthly visits for a minimum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age >= 18 years old
* BMI: < 30 and > 18
* Diagnosis of RA according to 2010 ACR/EULAR criteria and with a disease duration of at least 6 months since diagnosis
* Patient must present with active RA, characterized by at least 6 swollen joints out of 66 assessed and 6 tender joints out of 68 assessed and by the presence of synovitis (measured by ultrasound) in at least one of the 6 swollen joints
* C-reactive protein (CRP) level > 0.7 mg/dL or if the CRP level is between 0.3 mg/dL and 0.7 mg/dL (included) then patient must also present an ESR > 30mm/hr
* Patients must have received MTX treatment for at least 3 months and have been on a stable dose of MTX for at least 6 weeks prior to start of screening
* ACPA-positive RA patients
* Women must be postmenopausal (> 12 months without menses) or surgically sterile or using two effective contraception methods for at least 4 weeks prior to the randomization date and agree to continue contraception for the duration of their participation in the study (until the end of follow up period)
* Sexually active male patients must use a barrier method of contraception during the course of the study (and until the end of the follow up period)
* Patients must give written informed consent for study participation

Exclusion Criteria:

* A documented history of an autoimmune disease other than RA by ACR classification, or Sjögren syndrome
* Administration of cytotoxic drugs and immune suppressants (other than MTX) within 3 months prior to screening
* Previous multiple administrations of any biological DMARD or targeted synthetic DMARD
* Known primary immunodeficiency
* Pregnant or breastfeeding women
* Suspicion of active or latent tuberculosis
* HIV, HCV, HBV infection
* Infection reported during screening not recovered 72h prior to first dose
* History of anaphylactic reactions to any protein therapeutics or excipients
* Any history of malignancy, excluding cured basal or squamous cell carcinoma of the skin, or cervical in situ carcinoma
* Clinically significant cardiac disease requiring medication, such as congestive heart failure, unstable angina, myocardial infarction within 6 months prior to randomization
* Moderate to severe renal insufficiency, clinically relevant liver function test abnormalities or pancytopenia
* Major psychiatric or neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, causality and outcomes of Adverse Events (AEs) | From screening up to 24 weeks after first treatment administration
  Incidence, severity, causality and outcomes of Adverse Events (AEs) (serious and non-serious), with particular attention being paid to infusion-related reactions and infections
Withdrawal for safety reasons | From randomization up to 24 weeks after first treatment administration
Evolution of laboratory parameters | From screening up to 24 weeks after first treatment administration
Level of potential circulating antibodies against NI-0101 | From screening up to 24 weeks after first treatment administration
  Level of potential circulating antibodies against NI-0101 to determine immunogenicity; i.e. the development of anti-drug antibodies (ADA).
Levels of CRP | From screening up to 24 weeks after first treatment administration
  Levels of C-Reactive protein (CRP)
Levels of inflammatory cytokines/chemokines | From screening up to 24 weeks after first treatment administration
  IL-6, TNFa, IP-10, MCP-1, sICAM, CXCL13
DAS28 CRP | From screening to 24 weeks after first treatment administration
  Measure of Disease Activity Scores (DAS) for Rheumatism in 28 tender or swollen joints and C-Reactive protein (CRP) - DAS28-CRP
ACR criteria | From randomization to 24 weeks after first treatment administration
  Proportion of patients achieving American College of Rheumatology Criteria (ACR20, ACR50 and ACR70)
Proportion of patient achieving remission | From randomization to 24 weeks after first treatment administration
  Proportion of patient achieving remission (defined as DAS28 < 2.6)
EULAR response | From randomization to 24 weeks after first treatment administration
  Proportion of patients achieving European League Against Rheumatism (EULAR) response criteria - good, moderate and no response
Joint Count | From screening to 24 weeks after first treatment administration
  Mean number of Tender Joint Count/Swollen Joint Count.
SDAI score | From randomization to 24 weeks after first treatment administration
  Mean improvement from baseline in Simplified Disease Activity Index (SDAI) score
HAQ-DI score | From randomization to 24 weeks after first treatment administration
  Mean improvement from baseline in the Health Assessment Questionnaire without Disability Index (HAQ-DI) score
SF-36 score | from randomization to 24 weeks after first treatment administration
  Mean improvement from baseline in 36-Item Short-Form Health Survey (SF-36) score
DAS28-ESR | From screening to 24 weeks after first treatment administration
  Measure of Disease Activity Scores (DAS) for Rheumatism in 28 tender or swollen joints and Erythrocyte Sedimentation Rate (ESR) levels - DAS28-ESR
CDAI score | From randomization to 24 weeks after first treatment administration
  Mean improvement from baseline in Clinical Disease Activity Index (CDAI) score scores
Exploratory PK analysis - Cmax | From randomization to 24 weeks after first treatment administration
  Peak drug plasma concentration (Cmax)
Exploratory PK analysis - Tmax | From screening up to 24 weeks after first treatment administration
  Time when plasma concentration is at peak (Tmax)
Exploratory PK analysis - Ctrough | From randomization to 24 weeks after first treatment administration
  Plasma drug concentration immediately prior next dosing (Ctrough)
Exploratory PK analysis - AUC | From randomization to 24 weeks after first treatment administration
  Area under the plasma concentration versus time curve (AUC)
Exploratory PK analysis - CL | From randomization to 24 weeks after first treatment administration
  Systemic drug clearance (CL)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Choy, MD, Principal Investigator — Institute of Infection and Immunity, Cardiff University School of Medicine
Locations (19):
- Clinic for internal medicine with centre for dialysis, Mostar, Bosnia and Herzegovina
- Bulgaria (4):
  - Multi-profile Hospital for Active Treatment "Trimontsium", Plovdiv
  - University Multiprofile Hospital for Active Treatment "Kaspela", Plovdiv
  - Multiprofile Hospital for Active Treatment - Shumen AD, Shumen
  - University Multiprofile Hospital for Active TreatmenT "St. Ivan Rilski", Sofia
- Georgia (6):
  - ARENSIA Phase I Unit at the Research Institute of Clinical Medicine, Tbilisi
  - High Technology Medical Center; University clinic, Tbilisi
  - Emergency Cardiology Center by Acad. G.Chapidze, Tbilisi
  - Insitute of Clinical Cardiology, Tbilisi
  - Tbilisi Central Hospital, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- CRU Hungary Ltd, Miskolc, Hungary
- Republican Clinical Hospital, ARENSIA Phase I unit, Chisinau, Moldova
- Poland (2):
  - Centrum Miriada, Bialystok
  - Zespól Poradni Specjalistycznych REUMED, Lublin
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Special Hospital for Rheumatic Diseases "Novi Sad", Novi Sad
  - General Hospital "Djordje Joanovic", Zrenjanin